CLINICAL TRIAL: NCT01476241
Title: Percutaneous Endoscopic Gastrostomy Tube Placement by Otorhinolaryngologist: a Single Institution Experience
Brief Title: Percutaneous Endoscopic Gastrostomy Tube Placement by Otorhinolaryngologist
Status: Completed | Type: Observational
Sponsor: University of Helsinki (Other)
Responsible Party: Principal Investigator, Leif Back, Dr, University of Helsinki
Other Study IDs: PEG and ENT
Record Dates: First submitted 2011-11-15; First posted 2011-11-22 (Estimated); Last update posted 2011-11-22 (Estimated); Status verified 2011-11

CONDITIONS: Dysphagia
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- EarNoseThroatGroup: a cohort of patients that had undergone PEG tube placement from October 2008 until October 2010 at the Department of Otorhinolaryngology - Head and Neck Surgery
  Interventions: Procedure: PEG tube placement
- SurgeryGroup: a historic cohort group of patients with the PEG tube placed in the Department of Surgery from September 2005 until September 2009
  Interventions: Procedure: PEG tube placement

INTERVENTIONS:
Procedure: PEG tube placement — Percutaneous endoscopic gastrostomy
  Other Names: A) = EarNoseThroatGroup; B) = SurgeryGroup

SUMMARY:
The investigators main endpoint was focused on the analysis of the type, rate and the impact of different clinical parameters on the complications of the PEG tube placements performed at the Department of Otorhinolaryngology - Head and Neck Surgery since October 2008. In addition, the investigators aimed to compare the results with a historic cohort patient group (September 2005 - October 2008) sent to the Department of Surgery for PEG tube placement in order to evaluate the results of the changed routine.

DETAILED DESCRIPTION:
We retrospectively reviewed a cohort of patients that had undergone PEG tube placement from October 2008 until October 2010 at the Department of Otorhinolaryngology - Head and Neck Surgery, Helsinki University Central Hospital (HUCH), Helsinki, Finland, with a health care district currently including approximately 1.5 million inhabitants. Hospital surgical and discharge registries were used to identify the patients. Medical records were studied and details collected on the patients' age, sex, preoperative condition, preoperative laboratory parameters, coexisting medical diagnoses (Charlson Comorbidity Index, CCI (Hall 2004)), indication and date for PEG tube placement, complications, the time of PEG use, follow-up time, and clinical status at last follow up. The study period was aimed to run from PEG tube placement to the last clinical evaluation (minimum 12 months) or the time of death. These results were compared with those from a historic cohort group of patients with the PEG tube placed in the Department of Surgery, HUCH, Helsinki, Finland from September 2005 until October 2008.

ELIGIBILITY:
Inclusion Criteria:

* ENT patient with PEG tube placement

Exclusion Criteria:

* electrolyte imbalance
* coagulation imbalance
* morbid obesity (BMI > 40 kg/m2)
* large volume ascites
* previous gastrectomy
* sepsis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that had undergone PEG tube placement in a tertiary care center.
Sampling Method: Non-Probability Sample
Enrollment: 292 (Actual)
Dates: Start 2005-09; Primary Completion 2010-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Complications and mortality | 12 months follow-up time
  Complication
  * Minor
  * Major
  Mortality
  * Procedure related
  * < 7 days
  * 7-30 days
  * 30 days
  * Overall

CONTACTS AND LOCATIONS:
Overall Officials: Leif JJ Bäck, MD PhD, Principal Investigator — Dept of Otorhinolaryngology - Head and Neck Surgery, Helsinki University Central Hospital and University of Helsinki, Finland
Locations (1):
- Dept of Otorhinolaryngology - Head and Neck Surgery, Helsinki, Finland

REFERENCES:
- See also: Dept of Otorhinolaryngology - Head and Neck Surgery — http://www.hus.fi